CLINICAL TRIAL: NCT02197546
Title: Acupuncture Reduces Pain and Autonomous Distress During Injection of Local Anaesthetic in Children - a Randomised Crossover Investigation
Brief Title: Acupuncture for Pain During Injection of Local Anaesthetic
Acronym: AcuDent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BB 57/10; BB 57/10 (Other: BB 57/10)
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Pain; Distress; Satisfaction
Keywords: Injection pain; local anesthesia; acupuncture
MeSH Terms: conditions — Pain; Personal Satisfaction | interventions — Acupuncture Therapy; Acupressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- acupuncture plus local anesthesia (Other): Bilateral acupuncture with 1.5 mm long indwelling fixed needles
  Interventions: Other: Acupuncture & acupressure
- Local anesthesia alone (No Intervention): Standard therapy - local anesthesia alone without acupuncture

INTERVENTIONS:
Other: Acupuncture & acupressure — Bilateral acupuncture with indwelling fixed needles 1.5 mm length with subsequent acupressure by the parents
  Arms: acupuncture plus local anesthesia

SUMMARY:
Stimulation of acupoint LI4 has been shown to result in analgesic effects in patients experiencing acute pain. We aimed to determine whether LI4 acupuncture could reduce pain and distress in children receiving an injection of a local anaesthetic (LA). Children scheduled for dental treatment using local anesthesia as a standard treatment, received bilateral acupuncture at LI4 using indwelling fixed needles. During the treatment, the parents of the patients stimulated the needles by massage. Two different treatment regimes were compared: a standardized LA injection given 5 minutes after acupuncture, and an LA injection without acupuncture. The order of treatment was randomised, with the two treatments performed on different days. Pain intensity during LA injection, assessed by the patient with the Verbal Rating Scale or Faces Pain Scale (0-10), was used as the primary endpoint. Parent- and dentist-assessed pain intensity and agitation, heart rate, and the patients' satisfaction with the received therapy were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* children with an American Society of Anesthesiologists (ASA) physical status of I or II
* scheduled for at least two dental treatments for caries requiring local anaesthesia

Exclusion Criteria:

* history of analgesic medication, psychiatric disease, or local or systemic infection
* necessity to change their treatment schedule

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
pain intensity | 3 time points during one day of investigation

SECONDARY OUTCOMES:
pain intensity assessed by the parents and by physicians | 4 time points during one day of investigation

OTHER OUTCOMES:
heart rate | 5 time points during one days of investigation

CONTACTS AND LOCATIONS:
Overall Officials: Christian Splieth, MD, PhD, Study Chair — University Medicine of Greifswald
Locations (1):
- University Medicine of Greifswald, Greifswald, Germany